CLINICAL TRIAL: NCT04566185
Title: Evaluation of the Value of 18F-fluorodeoxyglucose Positron Emission Tomography (FDG PET) and Brain Perfusion Computed Tomography (CT Perfusion) for Predicting the Efficacy of Anti-angiogenic Therapy (Bevacizumab) in Patients With Recurrent Glioblastoma
Brief Title: Evaluation of the Predictive Value of 18F-fluorodeoxyglucose Positron Emission Tomography and Brain Perfusion Computed Tomography for the Efficacy of Anti-angiogenic Therapy (Bevacizumab) in Recurrent Glioblastoma
Acronym: EVA DOPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NIMAO/2018-03/LC-01
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with recurrent glioblastoma (Experimental)
  Interventions: Other: FDG PET; Other: CT scan; Other: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Other: FDG PET — IV application of F Dopa, 2 MBq per Kg, with a scout view (angle of view 90 °, 120 kV, 30 mAs), then an X-ray scan is performed for the attenuation correction ( 120 kV - 5mAs - pitch 0.531 - thickness // increment: 3.75mm//3.27mm -QAC filter - DFOV 25).
  PET acquisition: static in 3D mode for 20 minutes, 8 minutes after the injection of 18 F Dopa, the axial field of view is 25, the matrix in 256 x 256. After OSEM reconstruction 6 iterations and 24 subsets, with correction of attenuation and diffusion, then Gaussian filter of frequency 4, 47 contiguous axial sections of 3.26 mm are obtained.
Other: CT scan — Localization propeller without injection: 120kV - mA regulation (Noise Index 15) - pitch 0.969 - thickness // increment: 5mm // 5mm - Soft filter - Asir 60% - DFOV 25.
  Acquisition begins 5 seconds after the start of the injection of 60 ml of contrast product (VISIPAQUE) at 4 cc / second without (acquisition characteristics: 80 kV - 100 mAs -- thickness: 5mm // 8 images / rotation - STD filter - Asir 50% display field of view (DFOV) 25 - phase1: 5s then phase2 15s).
  Diagnostic quality CT: 120kV - Regulation of mA (Noise Index 15) - pitch 0.531 - thickness // increment: 1.25 // 0.625mm - Soft filter - Asir 60% - DFOV 25.
Other: Magnetic resonance imaging (MRI) — If the examination is performed on the SIEMENS SKYRA 3T device: 32 channel head coil antenna, if on the PHILIPPS INGENIA 1.5 T device: DStream HeadSpine Coil antenna.
  The sequence begins with an axial, coronal and sagittal "Survey" topogram, lasting 1 minute.
  Then axial sequence T1, Axial T2 *, Axial cerebral perfusion (Injection of gadolinium (0.1 mmol / kg, 5 cc / second), coronal T2, Axial T2 Flair, Axial DWI b100, Axial 3D T1 gadolinium

SUMMARY:
In this pilot study, the study evaluators will evaluate the ability of positron emission tomography (PET) with 18F-fluorodeoxyglucose (FDG PET) and the computed tomography (CT) perfusion scanner, individually and combined, to predict the effectiveness of anti-angiogenic treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient has an WHO score ≤ 3
* The patient's estimated life expectancy is more than 3 months.
* Patient with histologically proven diagnosis of glioblastoma.
* Patient presenting with tumor progression on morphological MRI confirmed by a multidisciplinary committee.
* Patient with a unilateral supratentorial target lesion upon inclusion to establish a tumor region of interest (ROI) zone and an equivalent ROI zone in contralateral healthy tissue.
* Patient progressing after radiotherapy and at least one line of chemotherapy with TEMODAL
* Patient in whom treatment with Bevacizumab monotherapy has been validated by a multidisciplinary committee.

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Pregnant or breast feeding patients
* Hypersensitivity to iodinated contrast media and creatinine clearance less than 60 ml / minute.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Categorization of patients as responders or non-responders to treatment | 2 months
  Measured by MRI according to Response Assessment in Neuro-Oncology (RANO) criteria: Complete response/Partial response/stable/progression

SECONDARY OUTCOMES:
Metabolic Tumor Volume | Day 0
  FDG PET
Metabolic Tumor Volume | Day 14
  FDG PET
Fixation Index | Day 0
  Maximum standard uptake value (SUV) and average SUV of the lesion divided by maximum SUV and average SUV of the striata
Fixation Index | Day 14
  Maximum standard uptake value (SUV) and average SUV of the lesion divided by maximum SUV and average SUV of the striata
permeability-surface area product | Day 0
  CT scan
permeability-surface area product | Day 14
  CT scan
cerebral blood flow | Day 0
  CT scan
cerebral blood flow | Day 14
  CT scan
Normalized permeability-surface area product to healthy brain | Day 0
  CT scan
Normalized permeability-surface area product to healthy brain | Day 14
  CT scan
Normalized cerebral blood flow to healthy brain | Day 0
  CT scan
Normalized cerebral blood flow to healthy brain | Day 14
  CT scan
Inter-rater reproducibility of FDG PET | End of study (September 2022)
  LIN intraclass correlation coefficient
Inter-rater reproducibility of CT scan | End of study (September 2022)
  LIN intraclass correlation coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Collombier, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France